CLINICAL TRIAL: NCT01194232
Title: Randomized Controlled Study of Sildenafil in Children and Young Adults With Mild to Moderate Cystic Fibrosis Lung Disease
Brief Title: Sildenafil Trial in Children and Young Adults With CF
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding, MedWatch change to study drug
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-2067
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Cystic Fibrosis With Mild to Moderate Lung Disease; CMRI of Lung Perfusion; Lung Perfusion; Lung Vascularization
Keywords: Cystic Fibrosis; CF; CMRI; vascularization; perfusion
MeSH Terms: conditions — Cystic Fibrosis; Neovascularization, Pathologic | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sildenafil (Experimental): 15 subjects will receive 8 week course of Sildenafil administered at a dose of 20 mg per dose three times per day.
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — 8 week course of Sildenafil administered at a dose of 1 mg / Kg three times a day with a maximum dose of 20 mg per dose.

SUMMARY:
Cystic Fibrosis (CF), the most common inherited disease in Caucasians, is characterized by chronic pulmonary inflammation and progressive loss of gas exchange units that eventually results in respiratory failure. There is strong evidence that, in CF, abnormally low perfusion carries a high risk of death independent from the presence of pulmonary hypertension. However, the evolution of pulmonary vascular disease in CF and how it might contribute to the rate of decline in lung function is not known. Our knowledge remains limited to the results of old observational studies which concluded that the major causes of pulmonary vascular remodeling and hypertension in CF are hypoxic respiratory failure and destruction of lung tissue. Our recent data obtained by state-of-the-art Magnetic Resonance Imaging (MRI) of the pulmonary circulation, challenges the existing paradigm. We demonstrate that in the absence of hypoxia, significant changes in pulmonary perfusion and in surrogate measures of vascular resistance as well as in collateral blood flow begin early in the course of CF. Newly developed therapeutics have altered dramatically the course of patients suffering from pulmonary vascular disease. Through this 8 week trial, we will examine by Magnetic Resonance Imaging the effect of Sildenafil on pulmonary perfusion and systemic vascularization of the lungs in subjects with mild to moderate disease.

ELIGIBILITY:
Inclusion Criteria

Research subjects must meet the following inclusion criteria:

* Age 8 years to age 21 years
* Weight > 20kg
* Diagnosis of cystic fibrosis confirmed by a prior sweat chloride evaluation of > 60 mmol/liter or by two identified CFTR mutations on genetic analysis
* Able to perform acceptable and repeatable spirometry per American Thoracic Society/European Respiratory Society (ATS/ERS) joint consensus criteria.
* Have valid spirometry data for at least 3 years
* Must have mild to moderate lung disease (Mild lung disease will be defined as an FEV1%p of 80-99% predicted. Moderate lung disease will be defined as an FEV1%p of 60-79% predicted.)
* If under the age of 18, the subject must assent to participation in the study, and the subject's parent or guardian must be able to give written informed consent and comply with the requirements of the study protocol
* If 18 years of age or older, the subject must be able to give written parental permission and comply with the requirements of the study protocol
* For female subjects: negative serum pregnancy test and must be willing to use contraception during study participation
* Able to tolerate MRI without sedation
* Subjects who are on alternating monthly on/off cycles of inhaled antibiotics must be willing to be off of inhaled antibiotic therapy for one "on" cycle.
* Must be currently enrolled in CCHMC IRB#: 2008-0926
* Normal Vitamin K status (PT/IND, PIVKA, etc) at screening

Exclusion Criteria

Research subjects will be excluded from the study based on:

* History of CF-related liver disease with portal hypertension
* Currently smoking cigarettes or other tobacco products
* Use of daytime oxygen supplementation
* Previous organ transplantation
* Unstable or uncontrolled hypertension
* Ongoing use of oral corticosteroids
* For female subjects: pregnancy or lactation and unwillingness to use contraception during study participation
* Any hemodynamically significant congenital or acquired cardiac disease or significant cardiomyopathy, hematologic disease (i.e. hemoglobinopathies), or pulmonary disease associated with an increased risk of pulmonary perfusion defects or pulmonary hypertension other than as an outcome of CF
* History of renal and/or hepatic insufficiency, defined as cystatin-C level that exceeds normal range and a previous diagnosis of liver cirrhosis.
* History of uncontrolled asthma defined as oral steroid dependent
* History of hypersensitivity to gadolinium (Magnevist)
* Contraindications specific to MRI including a history of claustrophobia, cardiac pacemaker, or other non-MRI compatible surgical implants (This includes neuro-stimulators containing electrical circuitry, or which generate electrical signals and/or have moving metal parts, and metal orthopedic pins or plates. The research coordinator and/or the MRI technologist will screen all subjects using the standard checklist of medical history and safety questions used by the Radiology Department in routine clinical scans.)
* Daily use of montelukast and ibuprofen
* Use of nitrate medicines or other drugs known to have unsafe interactions with Sildenafil
* Known allergy to Sildenafil
* Inability to comply with study procedures
* History of the following:

  1. Tinnitus or hearing impairment
  2. CF exacerbation within the preceding two months
  3. Ulcer, severe gastritis, or prior GI bleed
  4. Recurrent epistaxis
  5. Diabetes or abnormal OGTT (risk of retinal hemorrhage with sildenafil is highest in diabetics)

Laboratory Exclusion Criteria for research subjects (based on history or blood work before first MRI):

* Positive sputum, epiglottic, or bronchoalveolar lavage culture for Mycobacterium abscessus during the 2 years prior to enrollment
* A positive serum pregnancy test
* Serum creatinine > two times the upper limit of normal for age
* A serum Cystatin C < 60 ml/min/1.73m2
* Vitamin K outside of normal range

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Increase pulmonary perfusion | 8 week visit
  • Increase of pulmonary perfusion by a minimum of 15% as measured by gadolinium contrast MRI with segmental perfusion and scored on a continuous scale;

SECONDARY OUTCOMES:
Improved lung function | 8 weeks
  • Improved exercise performance as measured by the following variables:
  * Ventilatory equivalent of O2 and CO2 (VEO2 and VECO2)
  * Maximum oxygen consumption (VO2 max)